CLINICAL TRIAL: NCT00515398
Title: A Multicenter Study to Evaluate and Characterize the Effects of Pharmacological Chaperones in Cell Lines Derived From Blood and Skin Samples From Patients With Pompe Disease
Brief Title: A Study to Evaluate the Effects of Pharmacological Chaperones in Cells From Patients With Pompe Disease
Status: Completed | Type: Observational
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Irina Kline, Medical Director, Amicus Therapeutics
Other Study IDs: POM-CL-001
Record Dates: First submitted 2007-08-10; First posted 2007-08-13 (Estimated); Last update posted 2008-06-05 (Estimated); Status verified 2008-06

CONDITIONS: Pompe Disease; Glycogen Storage Disease Type II
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — White blood cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Group 1 (all subjects)
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Ex vivo administration of AT2220

SUMMARY:
The purpose of this study is to see how molecules called pharmacological chaperones affect the cells of patients with Pompe disease. The study will last 1 or 2 visits which will include a blood collection, urine collection, and two skin biopsies. Information will also be collected from the medical records about disease history and diagnosis. Patients will not receive any study medication.

DETAILED DESCRIPTION:
The study is designed to evaluate the response of cell lines derived from blood and skin tissue from Pompe patients to pharmacological chaperones. Samples of blood and skin tissue will be obtained to make cell lines that will be used to test pharmacological chaperones. The study will include patients with early and late-onset Pompe disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any age
* Confirmed diagnosis of Pompe disease (early or late-onset)
* Clinically stable
* Written informed consent by subject or legal representative

Exclusion Criteria:

* Other significant disease or otherwise unsuitable for the study, as determined by the investigator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Pompe disease
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-08; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
To evaluate and characterize the effects of pharmacological chaperones on enzyme activity and other markers of disease in cell lines derived from patients with Pompe disease | 1 week

SECONDARY OUTCOMES:
To study biomarkers associated with Pompe Disease and study the correlation between biomarkers and clinical disease state of patients with Pompe disease | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Irina Kline, MD, Study Director — Amicus Therapeutics
Locations (4):
- United States (4):
  - University of Florida, Gainesville, Florida
  - Washington University, St Louis, Missouri
  - Center for Metabolic Disorders, Lake Success, New York
  - Duke University, Durham, North Carolina